CLINICAL TRIAL: NCT03119298
Title: Measuring Fear of Physical Activity in Patients With Heart Failure Using Questionnaires and Physiological Parameters
Brief Title: Measuring Fear of Physical Activity in Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Trier (Other)
Collaborators: Krankenhaus der Barmherzigen Brüder Trier (Other)
Responsible Party: Principal Investigator, Prof. Dr. Heike Spaderna, Professor of Health Psychology, University of Trier
Other Study IDs: 10784
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Chronic Heart Failure; Fear of Physical Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High-fear-of-physical-activity group: Group members with high fear of physical activity
- Low-fear-of-physical-activity group: Group members with low fear of physical activity
- Control group: Healthy subjects matched for age and sex

SUMMARY:
The study's aims are twofold: First, to examine physiological correlates of fear of physical activity (PA) and second, to examine correlates between fear of PA and interoceptive abilities in patients with chronic heart failure and healthy persons. Patients' fear of PA will be assessed via the "Fear of Activity in Situations - Heart Failure" (FActS-HF) questionnaire. The patient group will be split into two subgroups: One with high fear of PA and the second with low fear of PA based on FActS-HF scores. Fear of PA will be assessed via an adapted version of FActS-HF in a sample of healthy persons (control group). Each member of the high-fear-of-PA group will be individually age- and sex-matched with one member of the low-fear-of-PA group and control group. The participants of all three groups undergo the same experimental trials.

Aim 1: The "startle paradigm" will be used to investigate the physiological component of fear of PA. The startle paradigm is based on empirical observations that the startle reflex is larger after the priming with unpleasant stimuli and inhibited after the priming with pleasant stimuli. The participants will be primed with various words including those words associated with physical activity that are expected to be unpleasant in patients with high fear of PA. The startle reflex will be triggered by air puffs on the eyes (startle probes) and measured via facial electromyography (EMG). We assume that startle responses primed with PA related words are stronger in patients with high fear of PA compared to the other groups.

Aim 2: Interoceptive accuracy will be assessed via the "Schandry test" and interoceptive awareness will be assessed via the "Multidimensional Assessment of Interoceptive Awareness" (MAIA) questionnaire. During the Schandry test the participants will be instructed to subjectively count their heart rate without any aid or tools. The heart rate will be objectively measured at the same time via ECG. A high congruence of the objective and subjective results indicates a high interoception ability, and is assumed to be correlated with fear of physical activity. Additionally, we expect the MAIA and FActS scores to be correlated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Heart Failure stage B or C (Hunt et al., 2005), or: New York Heart Failure classification II to IIIb

  1. Systolic dysfunction: left ventricular ejection fraction < 45% in the last 6 month
  2. Diastolic dysfunction: left ventricular ejection fraction >= 45% in the last 6 month

Exclusion Criteria:

* complex ventricular arrhythmias
* acute myocarditis
* symptomatic cardiac valve stenosis
* instable angina pectoris
* other severe diseases, that impair physical activity (e.g. advanced stages of cancer)
* insufficient language skills in German to answer the questionnaires
* insufficient cognitive skills to answer the questionnaires

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with diagnosed chronic heart failure of all underlying diagnoses. Patients have to be outpatients at time of study participation. They will be recruited in primary care clinics, and heart failure outpatient clinics in Germany. For the control group healthy volunteers without a chronic heart failure are recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Electromyography (EMG) magnitude (in µV) during startle probes | 30 minutes, one time point
  The startle reflex will be triggered by air puffs (startle probes) and its modulation in response to a set of verbal stimuli related to physical activity will be measured with the EMG during a time window of 30 minutes. Thereby physiological (EMG magnitude) correlates of fear of physical activity will be assessed.
Electrocardiography (ECG) measures of interbeat intervals and subjective counts of heart beats | 10 minutes, one time point
  Interoceptive accuracy will be assessed as the congruence of subjective heart beat counts and objectively measured ECG interbeat intervals (Schandry test) during specified time intervals.

SECONDARY OUTCOMES:
Scores on the Multidimensional Assessment of Interoceptive Awareness (MAIA) scale | 5 minutes, one time point
  The MAIA scale assesses the interoceptive awareness using the subscales emotional awareness, body listening, etc. Each item is rated on a continuous scale from 0 (never) to 5 (always). Sum scores of the subscales will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Heike Spaderna, Prof. Dr., Study Chair — Trier University
Locations (1):
- Department of Health Psychology, Trier University, Trier, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffmann JM, Hellwig S, Brandenburg VM, Spaderna H. Measuring Fear of Physical Activity in Patients with Heart Failure. Int J Behav Med. 2018 Jun;25(3):294-303. doi: 10.1007/s12529-017-9704-x. PMID 29230643